CLINICAL TRIAL: NCT02696109
Title: Cornerstone Program for Transition-Age Youth With Serious Mental Illness: Study Protocol for a Randomized Controlled Trial
Brief Title: Cornerstone Program for Transition-Age Youth Study Protocol for a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34-MH102525-01A1MRM; R34MH102525-01A1 (NIH)
Record Dates: First submitted 2015-12-10; First posted 2016-03-02 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2020-02

CONDITIONS: Depression; Stress Disorders, Post-traumatic; Bipolar Disorder
Keywords: Transition age youth; Mental health; Mental health services; Engagement
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Bipolar Disorder; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multimodal psychosocial intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cornerstone (Experimental): Participants in the experimental arm will be assigned a Transition Facilitator, a clinician with whom the client will meet one-on-one, and will be asked to attend once-a-week groups with other transition age youth. The groups will focus on issues relevant to successful transition to independent adulthood including stress and anger management and healthy relationships.
  Interventions: Behavioral: Cornerstone
- Treatment as Usual (Active Comparator): Participants in the TAU arm will be assigned to standard care at our partnering mental health agency. These clients are free to attend one-on-one counseling or any other services available at the clinic or elsewhere to address mental health challenges.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Treatment As Usual — Participants in the TAU arm will be assigned to standard care at our partnering mental health agency. These clients are free to attend one-on-one counseling or any other services available at the clinic or elsewhere to address mental health challenges.
  Arms: Treatment as Usual
Behavioral: Cornerstone — Participants in the experimental arm will be assigned a Transition Facilitator, a clinician with whom the client will meet one-on-one, and will be asked to attend once-a-week groups with other transition age youth. The groups will focus on issues relevant to successful transition to independent adulthood including stress and anger management and healthy relationships.
  Arms: Cornerstone

SUMMARY:
The purpose of this study is exploring a theoretically guided intervention, Cornerstone, which provides system 'boundary-spanning' services, including therapeutic services and mentorship, to transition-age youth with mental disorders. Cornerstone is designed to improve mental health service engagement and outcomes. The study uses a mixed methods approach to refine Cornerstone, and a hybrid design examining feasibility, acceptability, and preliminary impact with a randomized trial, alongside implementation.

DETAILED DESCRIPTION:
The goal of this RCT is to refine and examine the feasibility, acceptability and preliminary impact of a theoretically guided intervention that provides system 'boundary-spanning' services to improve mental health service use and outcomes for low-income, transition-age youth with mental disorders (TAYMD). Through the refinement and testing of this intervention, called Cornerstone, we aim to address mental health challenges as well as the practical obstacles, such as lack of education, housing, and employment, that impede successful transition to adulthood. Cornerstone addresses these challenges by providing a service delivery strategy that spans the transition from the child to the adult system.

Cornerstone centers on addressing three pressing problems: (1) the discontinuation, or at best fragmentation, of mental health care for TAYMD, (2) the lack of evidence-based interventions for TAYMD, and (3) the reality that promising practices for TAYMD, many of which Cornerstone builds upon, have not been tested with a sample that moves from child to adult services. Cornerstone deals with these problems in innovative ways at a time of transformation in health care. First, Cornerstone provides a 'boundary spanning case manager' (BSCM) across the transition. That is, rather than extending the age of service provision in the child system, we prioritize collaboration with the adult system and practical assistance to assure that the transition to developmentally and clinically appropriate adult services and independent adulthood happen at age 18. Second, Cornerstone incorporates an innovative form of social support, namely a recovery role model mentor (RRM) who is a decade older than TAYMD. The RRM co-facilitates weekly groups and provides important information and mentoring (i.e., modeling, connection) for TAYMD. Third, the development of Cornerstone is aligned with policy and practice transformation, particularly Affordable Care Act and New York State Medicaid Redesign, prioritizing coordinated, evidence-informed care for TAYMD, expansion of the workforce, and an emphasis on achieving functional outcomes and wellness.

The aims are 1) to develop and refine all manuals and protocols for Cornerstone, 2) to determine the feasibility, acceptability, and preliminary impact of 'Cornerstone' relative to treatment as usual (TAU) on mediating outcomes (e.g., stigma), service use, and improved mental health and functioning outcomes, and 3) to explore implementation of Cornerstone through individual and group interviews with key stakeholder partners on aspects of the transforming local, state and national service context (e.g., staffing, payment). As a multidisciplinary team of professionals on the local, state, and national level we are committed to bridging the science to service gap for youth transitioning to adulthood with mental health challenges. Using qualitative methods and an RCT, this study is the first to examine a true transition intervention. We believe mental health services research that focuses on the transition to adulthood with innovative service delivery strategies that span developmental silos will decrease the number of TAYMD with unmet mental health needs.

ELIGIBILITY:
Inclusion Criteria:

1. Be between ages 17 and 18 at time of enrollment in the study,
2. Diagnosed with a mental disorder, including those who are diagnosed with any other co-morbid disorders,

Exclusion Criteria:

1. Does not speak English
2. Documented IQ lower than 70

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Intention to Engage in Mental Health Services | Assessed at baseline
  Standardized scale developed and tested by Fishbein and colleagues
Intention to Engage in Mental Health Services | Assessed one year after baseline
  Standardized scale developed and tested by Fishbein and colleagues
Adherence to Medication | Assessed at baseline
  "How often in the past week have you taken your medication?" Response options are: 0 - never, 1 - rarely, 2 - sometimes, 3 - all of the time.
Treatment Continuation (or Dropout) | Assessed one year after baseline
  "Has the participant remained in services (or dropped out)?"

SECONDARY OUTCOMES:
Mental Health Recovery | Assessed at baseline
  Recovery Scale Short Form
Mental Health Recovery | Assessed one year after baseline
  Recovery Scale Short Form
Depression Symptoms | Assessed at baseline
  Center for Epidemiological Studies Depression Scale
Depression Symptoms | Assessed one year after baseline
  Center for Epidemiological Studies Depression Scale
Young Adult Employment and Education | Assessed at baseline
  Current employment and/or education
Young Adult Employment and Education | Assessed one year after baseline
  Current employment and/or education

OTHER OUTCOMES:
Cornerstone and Treatment as Usual Fidelity | Twice per group for one year
  6 items per session using Likert scale
Implementation Checklist | Bimonthly for one year
  Group facilitators will be asked questions related to implementation of the intervention, for example, barriers to young adult participation including time, transportation, staffing, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University Silver School of Social Work, New York, New York, United States

REFERENCES:
- [Derived] Cole AR, Adams DR, Ben-David S, Sapiro B, Villodas ML, Stanhope V, Jaccard J, Munson MR. Feasibility, Acceptability and Preliminary Implementation of the Cornerstone Program for Transition-Age Youth with Mental Health Conditions: A Mixed Methods Study. Adm Policy Ment Health. 2023 May;50(3):506-519. doi: 10.1007/s10488-023-01254-1. Epub 2023 Feb 4. PMID 36738385
- [Derived] Munson MR, Cole A, Stanhope V, Marcus SC, McKay M, Jaccard J, Ben-David S. Cornerstone program for transition-age youth with serious mental illness: study protocol for a randomized controlled trial. Trials. 2016 Nov 8;17(1):537. doi: 10.1186/s13063-016-1654-0. PMID 27825381